CLINICAL TRIAL: NCT03350191
Title: A PET/CT Study to Assess the Receptor Occupancy by SAR425899 After Repeat Dosing Using Radiolabelled Tracers for the Glucagon and GLP-1 Receptor in Overweight to Obese T2DM Patients
Brief Title: A Clinical Study to Investigate if SAR425899 Binds to the Liver and Pancreas in Overweight to Obese Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Antaros Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PDY15264; 2017-001789-23
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SAR425899

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAR425899 high dose (Experimental): Repeated once daily subcutaneous (SC) doses of SAR425899 administered over 20 days
  Interventions: Drug: SAR425899; Drug: [68Ga] Ga-DO3A-VS-Cys40-Tuna-2 (glucagon receptor tracer); Drug: [68Ga] Ga-DO3A-VS-Cys40-Exendin-4 (GLP-1 receptor tracer)
- SAR425899 low dose (Experimental): Repeated once daily SC doses of SAR425899 administered over 20 days
  Interventions: Drug: SAR425899; Drug: [68Ga] Ga-DO3A-VS-Cys40-Tuna-2 (glucagon receptor tracer); Drug: [68Ga] Ga-DO3A-VS-Cys40-Exendin-4 (GLP-1 receptor tracer)

INTERVENTIONS:
Drug: SAR425899 — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
Drug: [68Ga] Ga-DO3A-VS-Cys40-Tuna-2 (glucagon receptor tracer) — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
Drug: [68Ga] Ga-DO3A-VS-Cys40-Exendin-4 (GLP-1 receptor tracer) — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous

SUMMARY:
Primary Objectives:

To assess in overweight to obese T2DM patients:

* The glucagon receptor occupancy of SAR425899 at two dose levels in the human liver with positron-emission tomography (PET) imaging using [68Ga]Ga-DO3A-VS-Cys40-Tuna-2 as a tracer compound.
* The GLP-1 receptor occupancy of SAR425899 at two dose levels in the human pancreas with PET imaging using [68Ga]Ga-DO3A-VS-Cys40-Exendin-4 as a tracer compound.
* Pharmacodynamic effects on fasting plasma glucose and biomarkers of lipid metabolism.
* Pharmacokinetic parameters for SAR425899 after repeated subcutaneous (SC) doses in plasma.
* Safety and tolerability of SAR425899.

DETAILED DESCRIPTION:
Study duration is approximately 7 weeks with a 20 days treatment period.

ELIGIBILITY:
Inclusion criteria :

* Male and female patients, between 18 and 75 years of age, inclusive.
* Body weight between 60.0 and 120.0 kg, inclusive, body mass index between 28.0 and 38.0 kg/m2, inclusive.
* Diagnosis of type 2 diabetes mellitus for at least 1 year at the time of inclusion with stable metformin treatment prior to inclusion, with or without comorbidities related to type 2 diabetes mellitus.
* Fasting plasma glucose ≥ 90 mg/dL at screening.
* Glycosylated hemoglobin (HbA1c) ≥6.5% and ≤9 % at screening.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), urologic or infectious disease, hormonal active tumors (e.g. pheochromocytoma or insulinoma), or signs of acute illness that is not related to the metabolic status of the patient.
* Presence or history of drug hypersensitivity (including known allergic reactions associated with glucagon like peptide-1 (GLP-1) agonist treatment [exenatide, liraglutide, lixisenatide]), or allergic disease diagnosed and treated by a physician.
* Any intake of menopausal hormone replacement therapy, systemic corticosteroids, growth hormones, weight-loss drugs, antihyperlipidemic treatment, antihyperglycemic treatment [e.g., GLP-1 agonists, insulin, thiazolidinediones, dipeptidylpeptidase (DPP-IV) inhibitors, sodium/glucose cotransporter-2 (SGLT-2) inhibitors etc.]) during the treatment period and within 21 days before first dosing or within 5 times the elimination half-life or pharmacodynamic half-life of the medication (if known), with the exception of metformin, sulphonylureas (SU), standard antihypertensive treatment, statins and acetyl salicylic acid.
* Any condition possibly affecting gastric emptying or absorption from gastro-intestinal tract (e.g., gastric surgery, gastrectomy, bariatric surgery, malabsorption syndromes, gastroparesis, abdominal surgery other than appendectomy, hysterectomy, cholecystectomy and herniaplasty).
* Surgically treated obesity, bariatric surgery.
* Severe dyslipidemia with fasting triglycerides >450 mg/dL at screening.
* Severe hypoglycemia resulting in seizure/unconsciousness/coma or hospitalization for diabetic ketoacidosis in the last 3 months before screening.
* Persistent hyperglycemia not adequately controlled by metformin, SUs and/or diet/exercise.
* Diagnosed diabetic neuropathy, retinopathy, nephropathy or renal impairment (GFR <60 mL/min; estimate after Cockcroft-Gault) at screening.
* Unstable hypo- or hyperthyroidism (as assessed by TSH) at screening.
* History of pancreatitis or pancreatectomy.
* Amylase and/or lipase > 2 upper limit of normal (ULN) at screening.
* Personal history or family history of medullary thyroid cancer or a genetic condition that predisposes to medullary thyroid cancer.
* Elevated basal calcitonin (≥20 pg/mL / 5.9 pmol/L) at screening.
* Known past or present diseases or disorders of any target organ (liver, pancreas, spleen).
* Medical positron emitting tomography (PET), single photon emission computer tomography (SPECT), abdominal or thoracic computer tomography (CT) examination during the previous 12 months' time period.
* Claustrophobia.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Glucagon receptor occupancy | Day 1 and Day 20
  Change of glucagon receptor tracer binding in the liver with SAR425899 between Day 1 and Day 20

SECONDARY OUTCOMES:
GLP-1 receptor occupancy | Day 1 and Day 17
  Change of GLP-1 receptor tracer binding in the pancreas with SAR425899 between Day 1 and Day 17
Adverse events | Up to 27 days
  Number of adverse events in patients under treatment with SAR425899
Pharmacokinetics | Day 20
  Assessment of SAR425899 maximum plasma concentration (Cmax)
Change in fasting plasma glucose (FPG) | Day 1 to Day 20
  Absolute change in FPG from baseline to Day 20
Change in ketone bodies | Day 1 to Day 20
  Absolute change in ketone bodies from baseline to Day 20
Change lipid biomarkers | Day 1 to Day 20
  Absolute change cholesterol from baseline to Day 20
Change in volume of distribution (Vt) in the liver | Day 1 and Day 20
  Change of glucagon receptor tracer Vt in the liver with SAR425899 between Day 1 and Day 20
Change in Vt in the pancreas | Day 1 and Day 17
  Change of GLP-1 receptor tracer Vt in the pancreas with SAR425899 between Day 1 and Day 17
Average standard uptake values (SUVs) of PET tracers in the liver and pancreas | Day 1, Day 17 and Day 20
  Average SUVs for glucagon and GLP-1 tracer in liver and pancreas
Pharmacokinetics | Day 20
  Assessment of SAR425899 time to reach Cmax ( tmax)
Pharmacokinetics | Day 20
  Assessment of SAR425899 area under the concentration versus time curve (AUC)
Pharmacokinetics | Day 20
  Assessment of SAR425899 terminal elimination half-life ( t1/2)
Pharmacokinetics | Day 20
  Assessment of SAR425899 total body clearance from the plasma (CL)
Change lipid biomarkers | Day 1 to Day 20
  Absolute change in free fatty acids from baseline to Day 20
Change lipid biomarkers | Day 1 to Day 20
  Absolute change in triglycerides from baseline to Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 7520001, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Eriksson O, Velikyan I, Haack T, Bossart M, Laitinen I, Larsen PJ, Berglund JE, Antoni G, Johansson L, Pierrou S, Tillner J, Wagner M. Glucagonlike Peptide-1 Receptor Imaging in Individuals with Type 2 Diabetes. J Nucl Med. 2022 May;63(5):794-800. doi: 10.2967/jnumed.121.262506. Epub 2021 Sep 9. PMID 34503957